CLINICAL TRIAL: NCT01960101
Title: Development of a Milk Product Substitution for Patients Suffering From Xerostomia Caused by Psychotropic Drugs and Comparison of Its Efficiency With the Use of Aequasyal (Oxidized Glycerol Triester)Spray.
Brief Title: Development of a Milk Product Substitution for Patients Suffering From Xerostomia Caused by Medication
Acronym: LactoXeros
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other); Centre Hospitalier Universitaire Dijon (Other); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Ecole Nationale de l'Industrie Laitière (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C12-58; 2012-A01686-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Xerostomia
Keywords: xerostomia; Saliva; iatrogenic oral dryness; antidepressants; mouth dryness; milk product
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactoxeros milk product (Experimental): Patient will take the milk product orally for 14 days as many times as needed per day(but not more than 6 times daily).
  Interventions: Other: LactoXeros
- Aequasyal (Other): Patients will take the oral spray for 14 days. The Aequasyal ® Oral Spray is a solution of oxidized glycerol triesters. The oral spray is applied by spraying on the inside of each cheek, 3-4 times per day. After each administration, users are instructed to gently spread the product around the mouth with the tongue. The Aequasyal ® Oral Spray is a Class I medical device, and is CE-marked.
  Interventions: Device: Aequasyal

INTERVENTIONS:
Other: LactoXeros
  Arms: Lactoxeros milk product
Device: Aequasyal
  Arms: Aequasyal

SUMMARY:
Dry mouth is in most cases due to iatrogenic causes, particularly drugs. The existing products such as saliva substitutes are often disappointing (bad taste, poor efficiency).

Our hypothesis has considered the "empirical" observations made by some patients with xerostomia who consumed milk products to relieve the dry mouth syndrome from which they suffered. With this clinical observation, a closer collaboration has been undertaken with research laboratories specialising in food and especially milk. Through its composition, the dairy product in itself provides relief for the patient, due both to its physical and biochemical properties, which could explain these observed improvements, and elements related to the phenomena of consumption of food as an alternative to medication. In the latter, hedonism takes on a role which has not been previously assessed. Initial work undertaken with the department of applied research at the National Dairy Industry School (ENIL) led to the prototyping of a new natural milk, which is the subject of this application for development, to qualify and adapt a product with a "health benefit" in patients suffering from xerostomia.

To further develop this project we will initiate a sequential clinical trial by groups of five ambulatory patients with xerostomia (patients taking antidepressants followed in psychiatry appointments). The clinical tests will be organised by the CIC with the psychiatric wards of the University Hospital of Besançon. Each group of 5 patients will test a similar product for 14 days. The information collected after a series of tests with a group of patients will be translated by changing the ENIL specifications to produce a new mini-series of products. This repetition will be carried out up to 3 times if necessary to help achieve a satisfactory product in terms of taste, texture and lubrication properties, which will then be tested in a randomized controlled cross-over study of the efficiency and acceptability of the new "LactoXeros" product versus a reference product (Aequasyal ®, Oxidized Glycerol Triester) on a group of 32 patients at the University hospital of Dijon.

A natural way to combat xerostomia at the interface of patient diet, such as we propose, could help improve quality of life for patients, minimize harmful effects (infection, decay) and promote adherence of patients to treatments which are responsible for xerostomia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients seen in the psychiatry department requiring the prescription of psychotropic drugs (antidepressants anxiolytics) for over 6 weeks
* Patients complaining of xerostomia
* Patients having not taken a palliative therapy against xerostomia for at least 2 weeks
* Patients having signed a free and informed consent form
* Patients affiliated to a social security system

Exclusion Criteria:

* Patients suffering from psychotic illness
* Patients suffering from Sjogren's syndrome
* Patients having been treated by radiation therapy for head or neck cancer
* Patients having stopped a palliative therapy against xerostomia for less than 2 weeks
* Patients under 18
* Pregnant or Breastfeeding women
* Incapacitated adults
* Patients placed under tutorship or curatorship
* Patients under judicial protection
* Patients suffering from milk allergy or lactose intolerance
* Patients allergic to curcumin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Mouth Dryness Score | Score measured at day 0, day 14, Day 21 and day 35
  The mouth dryness score will be evaluated using a visual analogical scale (scale increased from 0 to 10 cm). The value 0 refers to normal mouth dampness (absence of dry mouth symptoms) and value 10 represents "the worst imaginable" dry mouth symptoms. This score is specific, sensitive and reproducible

SECONDARY OUTCOMES:
Perception of other symptoms of dry mouth | Day 0, 14, 21 and 35
  difficulty chewing, swallowing and speaking, burning sensation will also be evaluated using a visual analogical scale ranging from 0 to 10 cm
Silness-Loe Index measuring dental plaque | Day 0, 14, 21 and 35
  The oral examination will be performed by a dentist. During the inspection, the Silness Loe plaque index will be measured. The appearance of the oral tissue (redness, dryness) will be assessed using an ordinal 4-point scale as follows: 0 = none, 1 mild, 2 = moderate, 3 = severe
Salivary flow | Day 0, 14, 21 and 35
  People will be asked to spit in a collector tube for 8 minutes (2 sessions of 4 minutes separated by a 5-minute break). The saliva will be weighed and the salivary flow will then be calculated in g/min.
Biochemical analysis of saliva | Day 0, 14, 21 and 35
  * Antioxidant power (trolox)
  * Relative quantity of MUC5B mucin
  * Amylase activity
  * Lipase activity
  * Protein concentration
  * Proteolytic activity
  * Lysozyme level
Analysis of the mouth coating effect | Day 0, 14, 21 and 35
  assessed by optical fiber spectrofluorimetry detecting curcumin, a food coloring agent, on the tongue
Release of the aroma compounds | Between day 7 and 14 OR between day 28 and day 35
  This will be done only once and only when patients will be taking the experimental milk product (not with the Aequasyal product).
  Atmospheric Pressure Ionization Mass Spectrometry (API-MS) will be used for the continuous analysis of the retro-nasal release of flavor (nosespace) when chewing a sample of the milk product.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Haffen, Prof., Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (2):
- France (2):
  - Service de psychatrie adultes, Besançon
  - Service de Psychiatrie Adultes, Dijon